CLINICAL TRIAL: NCT05511480
Title: Reshaping the Motor Engram - An Online Crowdsourcing Study.
Acronym: FORGET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Kirstin-Friederike Heise, PhD, Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 00118731
Record Dates: First submitted 2022-08-11; First posted 2022-08-23 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Interference on sequence 1 (Experimental): The interference intervention (session six) will be applied to one of the two previously learned sequences (temporal).
  Interventions: Behavioral: Interference through learning of a competing motor skill.
- Interference on sequence 2 (Experimental): The interference intervention (session six) will be applied to one of the two previously learned sequences (spatial).
  Interventions: Behavioral: Interference through learning of a competing motor skill.
- Interference on sequences 1 and 2 (Experimental): The interference intervention (session six) will be applied to both of the two previously learned sequences (temporal and spatial).
  Interventions: Behavioral: Interference through learning of a competing motor skill.
- No interference (Sham Comparator): The interference intervention (session six) will be applied.
  Interventions: Behavioral: No interference

INTERVENTIONS:
Behavioral: Interference through learning of a competing motor skill. — Interference through the learning of a competing motor skill.
  Arms: Interference on sequence 1; Interference on sequence 2; Interference on sequences 1 and 2
Behavioral: No interference — No interference through the continuation of learning same motor skill
  Arms: No interference

SUMMARY:
A critical point in learning and memory research is whether memories, once consolidated, remain unchanged or whether they continue to undergo plastic changes and remodeling. While previous research has focused on experimental destabilization during early stages of the memory life cycle, i.e., during encoding or early consolidation, experimental data that provides information about the effect of destabilization interventions on well-consolidated memories is still missing. This is particularly true for the procedural memory domain, such as learning a sensorimotor skill. This project is designed to characterize the effect of a single behavioral interference intervention on a previously consolidated sensorimotor skill in a large sample of healthy volunteers recruited through an online crowdsourcing platform. In a longitudinal design, participants will perform an implicit sequence learning task over five consecutive sessions, followed by an interference intervention in session six and a follow-up evaluation of the stability of the learned skill in session seven. The experimental design includes two levels of sequential information (spatial and temporal), which allows the testing of the specificity of the interference intervention. Behavioral performance throughout the experimental sessions is acquired via the manual input on the participants' computer keyboards and used to extract the learning rate and the interference effect (primary outcome).

ELIGIBILITY:
Inclusion Criteria:

* registered Amazon Mechanical Turk users (called 'workers')
* with >95% approval rate on all previous Amazon Mechanical Turk assignments
* location in North America or Europe
* ≥18 years of age
* not having participated in this experiment before

Exclusion Criteria:

• prior participation in this experiment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Immediate interference rate (change in performance precision) | six days
  Performance in the learning task is derived from the precision of timing of key presses relative to the occurrence and duration of visual cues presented on the computer screen. The interference rate is operationalized as the change in performance precision over time.
  The immediate interference effect is analyzed based on the change in performance from before (pre-interference) the interference intervention to directly after the interference intervention in session six (post-interference). This change is normalized to the performance at baseline (pre-interference session six) and computed as [(post-interference - pre-interference)/pre-interference*100].
Delayed interference rate (change in performance precision) | seven days
  The delayed interference rate is calculated in analogy to the immediate interference effects with a 24-hours latency of the post-interference measure. Delayed interference is analyzed based on the change in performance from before the interference intervention (pre-interference in session six) to 24 hours after the interference intervention in session seven (24hours post-interference). This change is normalized to the performance at baseline (pre-interference session six) and computed as [(24 hours post-interference - pre-interference)/pre-interference*100].

SECONDARY OUTCOMES:
Learning rate (change in performance precision) | five days
  Skill learning is defined based on the precision of timing of key presses relative to the occurrence and duration of visual cues presented on the computer screen. Skill learning is indexed by increased precision over time, operationalized as declining deviation of key on- and offsets from the timing of cue on- and offsets. Learning rate is the absolute change of precision over the learning phase of five days, which is expected to follow an asymptotic exponential function.

CONTACTS AND LOCATIONS:
Overall Officials: Kirstin-Friederike Heise, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code